CLINICAL TRIAL: NCT00854763
Title: Phase 4 Study on Olmesartan, an Angiotensin Receptor Blocker, on Ambulatory Blood Pressure Change, Vitamin D Levels and Urinary Sodium Excretion of Patients With Hypertension
Brief Title: Olmesartan on Ambulatory Blood Pressure Change
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: National Taiwan University Hospital, National Taiwan University Hospital
Other Study IDs: 20091036M
Record Dates: First submitted 2009-03-01; First posted 2009-03-03 (Estimated); Last update posted 2009-03-03 (Estimated); Status verified 2009-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — olmesartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hypertension
  Interventions: Drug: olmesartan

INTERVENTIONS:
Drug: olmesartan — olmesartan

SUMMARY:
We will conduct an open label, non-comparative, observational study to evaluate the efficacy, safety and tolerability of Olmesartan therapy in Taiwan patients with essential hypertension, and the primary objective is the change in the 24-hour mean systolic blood pressure from baseline to the day after post-treatment week-12 visit according to the ambulatory blood pressure monitoring.

DETAILED DESCRIPTION:
Vitamin D plays an important role for cardiac function and blood pressure regulation, and the serum 25(OH)D concentration change is an important indicator for Vitamin D nutritional status, and serum 1,25(OH)2D is an active hormone for biological actions. However, little is known about the change of vitamin D concentration was related to the usage of angiotensin receptor blocker among patients with hypertension.

We will conduct an open label, non-comparative, observational study to evaluate the efficacy, safety and tolerability of Olmesartan therapy in Taiwan patients with essential hypertension, and the primary objective is the change in the 24-hour mean systolic blood pressure from baseline to the day after post-treatment week-12 visit according to the ambulatory blood pressure monitoring. Our second endpoints included:

1. Change in the 24-hour mean diastolic blood pressure from baseline to the day after post-treatment week-12 visit
2. To evaluate the reduction in office blood pressure, including SeSBP and SeDPB, with Olmesartan 20mg therapy at 4,8,12 weeks (only for subjects with week-4, week-8 visit)
3. Control rate [% of patients] at 12weeks, defined by Defined as SBP less than 140mmHg and / or DBP less than 90mmHg or a reduction more than 10 mmHg for DBP and / or more than 20mmHg SBP versus baseline values
4. Biomarker assessment Vitamin D change from the baseline 24-hour urinary sodium excretion change from the baseline
5. To evaluate the efficacy and tolerability of Olmesartan 20mg at 12 weeks based on global assessment by the physicians and patients

The major aim of this proposal is to investigate the effect of angiotensin receptor blocker, Olmesartan, for a 12 weeks' treatment among patients with hypertension in the outpatient clinics in one hospital center. We set the blood pressure measured from ambulatory blood pressure monitor as the primary endpoint. Furthermore, we will test Vitamin D related concentrations and 24 hour urine sodium excretion change with the blood pressure change. We will recruit 200 patients with hypertension in this observational study and will evaluate the efficacy and safety issues among these patients. The specific aims of this proposal will include:

1. Test the improvement of blood pressure change in 24-hour blood pressure monitor by an angiotensin receptor blocker, Olmesartan, among hypertensive patients
2. Test the change of vitamin D concentrations and 24-hour urinary sodium excretion change after this angiotensin receptor blocker, Olmesartan, treatment
3. Test the association between blood pressure change and vitamin D-related measurements among the drug treatment, We hypothesize that the blood pressure change was related to the change of serum vitamin D concentration and also related to urinary sodium excretion change. .

The unique feature of this proposal includes a well-designed observational study with experienced clinicians and epidemiologists to conduct the study. Under the infrastructure in a tertiary hospital center, participant compliance, follow up, quality control and outcomes measurements can be assured and monitored under the guideline of good clinical practice. Furthermore, the investigators are the experts in vitamin D associated measurements and biomarkers studies and in clinical setting. This proposal will provide important scientific knowledge about the relationship among blood pressure change, vitamin D and urinary sodium excretion among hypertensive patients under 12 weeks' angiotensin receptor blocker treatment in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or over.
* naïve patients with Stage I** or Stage II** (JNC VII) essential hypertension or patients uncontrolled on current hypotensive drug therapy (in cuff BP>140/90mm Hg)
* All selected patients must give their written informed consent before recording their personal data

Exclusion Criteria:

* Subject with secondary form of hypertension
* Subject is being treated or with unstable condition for disease of myocardial infarction, clinically decompensated congestive heart failure, angina pectoris, sick sinus syndrome, second or third degree atrioventricular block
* Subject with history of hypertensive encephalopathy, grade 3 or 4 hypertensive retinopathy within 3 months before entering this trial
* Subjects with a cerebrovascular accident within 6 months before entering this trial
* Subject with auto-immune disease
* Subject with uncontrolled endocrine diseases, such as Hyperthyroidism, Hypothyroidism, Hypercorticism and Hypocorticism
* Subject with confirmed evidence of renal impairment (creatinine > 1.5 x upper limit of normal)
* Subject with hyperkalemia with serum potassium > 5.5 meq/L
* Subject with terminal stage of malignant disease
* Subject with substance abuse history
* Subject with gastrointestinal disease which can interfere the absorption of the oral medications
* Subject with any contraindication to the use of angiotensin II receptor blocker or calcium channel blocker
* Subject is pregnant or lactating
* Premenopausal subjects not taking reliable methods for contraceptives
* Subject with any other serious disease considered by the investigator not in the condition to enter the trial
* Subject is not able to comply to the protocol requirements
* Subject participated investigational drug trial within 3 months before entering this study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 patients with hypertension who received an angiotensin receptor antagonist, Olmesartan, for 12 weeks' treatment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-04

PRIMARY OUTCOMES:
The primary objective is the change in the 24-hour mean systolic blood pressure from baseline to the day after post-treatment week-12 visit according to the ambulatory blood pressure monitoring. | 12 weeks

SECONDARY OUTCOMES:
Change in the 24-hour mean diastolic blood pressure from baseline to the day after post-treatment week-12 visit | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kuo-Liong Chien, MD, PhD, Principal Investigator — Institute of Preventive Medicine, College of Public Health, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan